CLINICAL TRIAL: NCT02055391
Title: A Randomized Controlled Trial of a Novel Weight Loss Intervention for Obesity
Brief Title: A Weight Loss Trial for Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Edie Goldbacher, Principal Investigator, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F32DK083910 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Weight Loss (Active Comparator): State of the art behavioral weight loss treatment
  Interventions: Behavioral: Behavioral Weight Loss
- Enhanced Behavioral Weight Loss (Experimental): Combines behavioral weight loss skills with skills specifically targeting emotional eating.
  Interventions: Behavioral: Enhanced Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Behavioral Weight Loss — Weekly group meetings addressing behavioral weight loss skills including calorie counting, exercise, behavior modification, environmental changes, and coping with triggers.
  Arms: Behavioral Weight Loss
Behavioral: Enhanced Behavioral Weight Loss — Weekly group meetings that combine behavioral weight loss skills (calorie counting, exercise, behavior modification, environmental changes) with skills to decrease emotional eating by learning ways to manage and cope with emotions without eating.
  Arms: Enhanced Behavioral Weight Loss

SUMMARY:
The purpose of this study is to determine whether a new weight loss treatment which incorporates behavioral weight loss skills and skills for learning how to identify, manage, and cope with emotions helps with weight loss and emotional eating in people who are overweight and eat in response to emotions.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, free of diabetes, overweight and interested in losing weight, eat in response to emotions

Exclusion Criteria:

* Diabetes, any major medical or psychiatric condition that would compromise ability to participate, hypertension, current mental health treatment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
weight change | 12 weeks and 20 weeks

SECONDARY OUTCOMES:
changes in emotional eating | 12 weeks and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edie M Goldbacher, PhD, Principal Investigator — Universidad La Salle, Mexico
Locations (1):
- CORE, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Goldbacher E, La Grotte C, Komaroff E, Vander Veur S, Foster GD. An initial evaluation of a weight loss intervention for individuals who engage in emotional eating. J Behav Med. 2016 Feb;39(1):139-50. doi: 10.1007/s10865-015-9678-6. Epub 2015 Sep 4. PMID 26341357